CLINICAL TRIAL: NCT03961087
Title: Impact of Coenzyme Q10 and Meclofenoxate on Frequency and Severity of Hepatic Encephalopathy
Brief Title: Coenzyme Q10 and Meclofenoxate in Hepatic Encephalopathy
Acronym: EH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Shaaban Hanafy, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5501
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Hepatic Encephalopathy; Coenzyme Q10; Intellectual Functioning Disability
MeSH Terms: conditions — Hepatic Encephalopathy; Intellectual Disability | interventions — coenzyme Q10; Meclofenoxate

STUDY DESIGN:
Intervention Model Description: patients with liver cirrhosis and frequent hepatic encephalopathy (HE)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case group (Active Comparator): patients with liver cirrhosis and frequent hepatic encephalopathy received coenzyme Q10 and Meclofenoxate in addition to usual hepatic support
  Interventions: Drug: Coenzyme Q10; Drug: MECLOFENOXATE
- control group (No Intervention): patients with liver cirrhosis and frequent hepatic encephalopathy received usual hepatic support only

INTERVENTIONS:
Drug: Coenzyme Q10 — Coenzyme Q10 will be given twice
  Other Names: coQ10
  Arms: case group
Drug: MECLOFENOXATE — MECLOFENOXATE will be given as 500 mg once daily.
  Other Names: LUCIDREL
  Arms: case group

SUMMARY:
Hepatic encephalopathy is a syndrome occurs in patients with liver cirrhosis and is defined as neuropsychiatric abnormalities in patients with liver impairment, characterized by personality changes, intellectual impairment, and an impaired level of consciousness.

Coenzyme Q10 (CoQ10) is a necessary cofactor of the mitochondrial metabolism. It provides a High antioxidant and protective effects on age-related morbidities such as hypertension, heart failure and neurodegenerative diseases and hepatoprotective effects in drug related hepatic impairment.

Meclofenoxate is a cholinergic nootropic drug used clinically to improve memory, mental function and general cognition.

DETAILED DESCRIPTION:
Hepatic encephalopathy is a syndrome occurs in patients with liver cirrhosis and is defined as neuropsychiatric abnormalities in patients with liver impairment, characterized by personality changes, intellectual impairment, and an impaired level of consciousness. Hepatic encephalopathy is categorized into Type A hepatic encephalopathy associated with acute liver failure; Type B hepatic encephalopathy is associated with portal-systemic bypass and no intrinsic hepatocellular disease; Type C hepatic encephalopathy describes encephalopathy associated with Cirrhosis and portal hypertension; type C hepatic encephalopathy is, in turn, subcategorized as episodic, persistent, or minimal.

A number of theories had been postulated, it was proposed that hepatic encephalopathy is a disorder of astrocyte function which play a key role in the regulation of the blood-brain barrier, maintaining electrolyte homeostasis , a role in the detoxification of chemicals, including ammonia.

neurotoxic substances, including ammonia and manganese cause morphologic changes in the astrocytes leading to Alzheimer type II astrocytosis in cirrhosis.

Hepatic encephalopathy may be due to accumulated neurotoxic substances in the brain as short-chain fatty acids; mercaptans; false neurotransmitters, such as tyramine, octopamine, and beta-phenylethanolamines; manganese; ammonia; and gamma-aminobutyric acid (GABA).

Coenzyme Q10 (CoQ10) is a necessary cofactor of the mitochondrial metabolism. It provides a High antioxidant and protective effects on age-related morbidities such as hypertension, heart failure and neurodegenerative diseases and hepatoprotective effects in drug related hepatic impairment.

Meclofenoxate is a cholinergic nootropic drug used clinically to improve memory, mental function and general cognition.

ELIGIBILITY:
Inclusion Criteria:

* All the patients diagnosed as having liver cirrhosis Exclusion Criteria
* recent alcohol intake;
* Infection, recent antibiotic use or gastrointestinal bleeding;
* use of drugs affecting psychometric Performances like benzodiazepines, antiepileptics, psychotropic drugs
* History of shunt surgery or transjugular intrahepatic portosystemic shunt for portal hypertension;
* Electrolyte abnormalities
* Renal impairment or hepatorenal syndrome
* hepatocellular carcinoma;
* Severe medical co-morbidities that affect quality-of-life measurement as heart failure pulmonary or neurological insults.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
hepatic encephalopathy | 6 months
  Change in the number of episodes
health related quality of life | 6 months
  health related quality of life questionnaire
hepatic detoxifying function | 6 months
  reduction of serum ammonia

CONTACTS AND LOCATIONS:
Overall Officials: Amr S Hanafy, M.D, Principal Investigator — Assistant prof of medicine-Zagazig University
Locations (1):
- Amr Shaaban Hanafy, Zagazig, Alsharkia, Egypt